CLINICAL TRIAL: NCT06522776
Title: Effectiveness of Brief Remote Psychological Intervention for COVID-19 Survivors With Acute Kidney Injury and Their Informal Primary Caregivers
Brief Title: Remote Psychological Intervention for COVID-19 Survivors With AKI and Caregivers (REPICOV-AKI)
Acronym: REPICOV-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesus Rivero, MD (Other Government)
Responsible Party: Sponsor-Investigator, Jesus Rivero, MD, MD, Instituto Nacional de Enfermedades Respiratorias
Organization: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C34-21
Record Dates: First submitted 2024-07-24; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Anxiety; Depressive Symptoms; Acute Kidney Injury
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression; Acute Kidney Injury | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote cognitive behavioral therapy (Experimental): A single-case experimental design A-B with prospective follow-up. We used the Patient Health Questionnaire-9 (PHQ-9) and the General Anxiety Disorder Scale-7 (GAD-7) to screen for depressive and anxiety symptoms, one week later after hospital discharge. Those with moderate or severe symptoms received cognitive behavioral therapy (CBT) and were evaluated over time with the instruments and daily self-report of symptoms.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — The investigator adapted the manual of psychological intervention based on Cognitive Behavioral Therapy (CBT) which previously was validated in patients with chronic kidney disease. Patients received CBT using a model of six modules, with a time of 60 minutes for each weekly session. For each module, a skill acquisition criterion was used, to know if the participants were putting the techniques into practice in their daily lives and to know if it was pertinent to move on to the next module. Modules were adapted to the needs of each participant. In consequence, the number of sessions was different for each patient. All participants had a follow-up session one month after they finished the psychological therapy. Additionally, a daily self-record of symptoms perception and a short questionnaire on the usefulness of each technique used were sent daily to the participants via a phone text message.

SUMMARY:
The frequency of psychological conditions in recovered COVID-19 patients with Acute Kidney Injury (AKI) and their informal primary caregivers (IPC) is unknown; as well as the effects of psychological therapy in this population. The present study was initiated to determine the effectiveness of a brief remote psychological intervention (BRPI) to reduce anxious and depressive symptoms in survivors of AKI.

The investigator designed a single-case experimental design A-B with prospective follow-up. We used the Patient Health Questionnaire-9 (PHQ-9) and the General Anxiety Disorder Scale-7 (GAD-7) to screen for depressive and anxiety symptoms, one week later after hospital discharge. Those with moderate or severe symptoms received cognitive behavioral therapy (CBT) and were evaluated over time with the instruments and daily self-report of symptoms. The statistical analysis was conducted using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of severe COVID-19 who had AKI during hospitalization
* Informal primary caregivers

Exclusion Criteria:

* They did not accept to participate in the study
* They did not answer three attempted phone calls or text messages making it impossible to complete the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Anxious symptoms score for identifying changes in psychological behavior before and after to brief remote psychological intervention. | From the date of one week later after hospital discharge at the hospital until the date of the end intervention, in average one month
  Psychological behavior changes were evaluated by the anxious symptoms score (mild, moderate, and severe) using General Anxiety Disorder Scale-7 (GAD-7).
Depressive symptoms score for identifying changes in psychological behavior before and after to brief remote psychological intervention. | From the date of one week later after hospital discharge at the hospital until the date of the end intervention, in average one month
  Psychological behavior changes were evaluated by the depressive symptoms score (mild, moderate, and severe) using the Patient Health Questionnaire-9 (PHQ-9).

SECONDARY OUTCOMES:
General perception scale for identifying the utility of each technique used for the management of psychological symptoms. | From the date of one week later after hospital discharge at the hospital until the date of the end intervention, in average one month
  The utility of each technique used for the management of psychological symptoms was evaluated by the general perception scale using a short questionnaire with daily self-record of symptoms perception (0-10 scale).

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rivero, MD, Principal Investigator — INER
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No